CLINICAL TRIAL: NCT00653666
Title: Metabolic Consequences of CPT1A Deficiency in Alaska Native Children
Brief Title: Metabolic Consequences of CPT-1 Deficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Alaska Department of Health and Social Services (Unknown)
Responsible Party: Melanie Gillingham, PhD, Oregon Health & Science University
Organization: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: CTRC1029 (completed)
Record Dates: First submitted 2008-04-03; First posted 2008-04-07 (Estimated); Last update posted 2010-02-25 (Estimated); Status verified 2010-02

CONDITIONS: Carnitine Palmitoyl Transferase Type 1A (CPT1A) Deficiency
Keywords: CPT1A; steatosis; deficiency; metabolic; response; fasting
MeSH Terms: conditions — Fatty Liver; Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Medically supervised fasting — Metabolic fasting studies will be conducted over an 18-hour period or until blood glucose is < 40 mg/dl. If the YSI reading is 40 mg/dl or less, at any time during the study, then a blood sample will be collected, and the fast terminated by giving D25W IV and then feeding orally.

SUMMARY:
The purpose of this study is to learn more about how long children with CPT-1 deficiency can wait between meals without developing low blood sugar or symptoms of low blood sugar. The other purpose is to learn more about how much fat is stored in the liver of a child with CPT-1 deficiency.

DETAILED DESCRIPTION:
With the advent of enhanced screening (via tandem mass spectroscopy, MS/MS), the Northwest Regional Newborn Screening Program (NWRNSP) has identified a high incidence of carnitine palmitoyl transferase type 1A (CPT1A) deficiency in Alaska Native infants. Since October of 2003 approximately 80 Alaska Native infants have been identified with this condition; previously only 30 published cases were known worldwide. All of the infants are homozygous for a c.1436C-T sequence variant in the CPT1A gene, which results in the substitution of a leucine for proline at amino acid position 479 (P479L), and an approximately 80% reduction of CPT1A activity (non-classic CPT1A deficiency) (7). The clinical implications of this very restricted level of enzyme activity are not known. However, patients with more severe reductions of CPT1A activity (as the result of other mutations) are known to be at high risk for hypoketotic hypoglycemia, liver dysfunction, and sudden unexplained death (1). Hepatomegaly with micro- and macro-vesicular steatosis is also common (16). Currently the treatment of Alaska Native infants and children with CPT1A deficiency is based on data from patients with more severe forms of CPT1A deficiency and other fatty acid oxidation (FAO) disorders. Our ultimate goal is to establish evidence-based guidelines for treatment of the form of CPT1A deficiency prevalent in the Alaska Native population. This pilot study addresses two specific questions and will provide the first glimpse of the physiologic effects of homozygosity for the c.1436C-T sequence variant in the CPT1A gene. These data will aid in the development of strategies for clinical management that can be evaluated in future prospective studies, and provide preliminary data required for applications for NIH funding for more in-depth characterization of the clinical consequences of this condition.

ELIGIBILITY:
Inclusion Criteria:

* CPT-1 deficiency
* homozygous for the c.1436C-T sequence variant
* greater than 6 kg
* otherwise healthy
* siblings must be free of CPT-1 deficiency but heterozygous for c.1436C-T sequence variant and otherwise healthy

Exclusion Criteria:

* liver dysfunction
* diabetes
* renal disease
* metal plate in body

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2007-10; Primary Completion 2008-11 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
To compare body composition, liver and muscle lipid content, and liver function of Alaska Native children with CPT1A deficiency, with similar measures in their unaffected siblings. | February 2009

SECONDARY OUTCOMES:
To characterize the metabolic response of Alaska Native children with CPT1A deficiency to fasting, | February 2009

CONTACTS AND LOCATIONS:
Overall Officials: Melanie B. Gillingham, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Derived] Gillingham MB, Hirschfeld M, Lowe S, Matern D, Shoemaker J, Lambert WE, Koeller DM. Impaired fasting tolerance among Alaska native children with a common carnitine palmitoyltransferase 1A sequence variant. Mol Genet Metab. 2011 Nov;104(3):261-4. doi: 10.1016/j.ymgme.2011.06.017. Epub 2011 Jun 28. PMID 21763168